CLINICAL TRIAL: NCT02692365
Title: Exploratory Study to Determine Tissue Alterations of Advanced Hepatocellular Carcinoma Induced by Electromagnetic Waves of Low Energy Amplitude Modulated to Specific Frequencies During Imaging Study by MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sirio-Libanes (Other)
Responsible Party: Principal Investigator, Frederico Perego Costa, Doctor, Hospital Sirio-Libanes
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HSL 2015-75
Record Dates: First submitted 2015-09-10; First posted 2016-02-26 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Primary or Metastatic Tumor in the Liver Parenchyma
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; Hemodynamics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Calcium channels (Experimental): Magnetic Resonance assessment Hemodynamics + + infusion of manganese chloride
  Interventions: Procedure: Magnetic Resonance + hemodynamic + infusion of gadolinium
- Tumor perfusion (Experimental): Magnetic Resonance + hemodynamic + infusion of gadolinium
  Interventions: Procedure: Magnetic Resonance + hemodynamic + infusion of gadolinium

INTERVENTIONS:
Procedure: Magnetic Resonance + hemodynamic + infusion of gadolinium
  Other Names: Magnetic Resonance assessment Hemodynamics + + infusion of manganese chloride

SUMMARY:
This is an exploratory, national, single-center, open-label study, being conducted at the Institute of Education and Research of the Syrian-Lebanese Hospital in collaboration with the Radiology Institute, the Heart Institute of the Faculty of Medicine of São Paulo, Hospital São Paulo UNIFESP, and the Departments of Physics and Mathematics at the University of São Paulo in order to detect the presence of calcium flux change, tumor perfusion and electrical properties of tumor tissue when exposed to RF EMF AM by Cancer-frequency specific in patients with advanced HCC and correlate these findings with hemodynamic changes assessed by non-invasive hemodynamic measurements.

This study aims to demonstrate the presence of three mechanisms (hypothesis) that could be involved in the hemodynamic changes and the specific antitumor effect induced by exposure to RF EMF AM cancer-specific frequency. This study is not intended to study a therapeutic or diagnostic procedure. For this reason, will not be considered evolutionary clinical data during and after the intervention of the study.

ELIGIBILITY:
Inclusion Criteria:

All individuals selected for these studies should be in accordance with the following inclusion criteria:

* Patients must have a diagnosis of HCC.
* Presence of the primary or metastatic tumor at the time of the procedure, at least one (1) measurable lesion by RECIST criteria modified located in the hepatic parenchyma and size> 2 cm.
* Patients with AFP> 400 ng / ml and image feature not need histopathological confirmation. But in patients with active B virus serology, the value of AFP should be greater than 4000 ng / ml. The remaining patients should be histological confirmation of HCC.
* Patients may be in observation or presence of systemic or intra-hepatic treatment.
* Minimum age 18 years.
* be subjected to MRI study without need for sedation.

Exclusion Criteria:

* Individuals selected for this study will be excluded if they are in accordance with the following exclusion criteria:

  * can not suspend anti-hypertensive drugs or beta blockers for at least 48 hours or be pacemaker carriers or other implantable device.
  * Any restriction known to carry out study of magnetic resonance imaging.
  * menstrual delay, pregnant or breastfeeding.
  * Presence of metal artifacts or implants that can alter the reading of the magnetic signal or heat or move during the MRI procedure.
  * Prior allergic Event Knowledge gadolinium or manganese chloride solution.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Exploratory study for the determination of tissue changes of advanced hepatocellular carcinoma induced by electromagnetic waves amplitude modulated low energy specific frequencies during image MRIstudy. | 30 min
  Procedure 1 - calcium channel They will be provided for ten (10) patients allocated for this study. Patients will undergo a two (2) studies of MRI with a minimum interval of 7 days between the two studies.
  Day - 8: according to a study of MRI and hemodynamic evaluation Procedure 2 - tumor perfusion They will be provided for ten (10) patients allocated for this study. Patients will undergo a two (2) studies of MRI with a minimum interval of 7 days between the two studies.
  Day - 1: first study of MRI Day - 8: according to a study of MRI and hemodynamic evaluation Procedure 3 - electrical properties of the tumor and metabolomics Procedure 4 - static magnetic field exposure They will be provided for 20 (twenty) patients allocated for this study. Patients will not be subjected to MRI studies.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sírio-Libanês, São Paulo, São Paulo, Brazil